CLINICAL TRIAL: NCT00005787
Title: Ex Vivo Expanded Peripheral Blood Mononuclear Cells for the Elimination of Neutropenia Associated With High Dose Chemotherapy
Brief Title: Peripheral Stem Cell Transplantation to Prevent Neutropenia in Patients Receiving Chemotherapy for Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Per PI due to poor/inadequate accrual.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: NU 99Z1; NU-99Z1; NCI-G00-1734
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma; Neutropenia
Keywords: neutropenia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Neutropenia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Epoetin Alfa; Filgrastim; flt3 ligand protein; Stem Cell Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: epoetin alfa
Biological: filgrastim
Biological: recombinant flt3 ligand
Biological: recombinant interleukin-3
Biological: sargramostim
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill cancer cells. Treating the peripheral stem cells in the laboratory may improve the effectiveness of the transplant.

PURPOSE: Phase I trial to study the effectiveness of peripheral stem cell transplantation in patients who have relapsed or refractory non-Hodgkin's lymphoma and who will be treated with high-dose chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of ex vivo expanded peripheral blood mononuclear cells (EVE PBMNC) as a supplement to high-dose chemotherapy and conventional autograft in patients with relapsed or refractory non-Hodgkin's lymphoma.
* Compare the effect of EVE PBMNC on white blood cell, red blood cell, and platelet recovery in patients on this study vs historical controls, matched by protocol, disease status, and prior therapy.
* Determine the optimal duration of culture and time of harvest for the production of neutrophils in vivo.
* Determine the relationships between length of culture, immunophenotype, and clinical outcome.
* Determine the required numbers of white blood cell precursors for clinical efficacy.
* Assess the need for multiple transfusions of EVE PBMNC during the post-transplantation period.

OUTLINE: Autologous peripheral blood mononuclear cells (PBMNC) are harvested. Unselected PBMNC are cultured and expanded ex vivo in flt3 ligand, interleukin-3, filgrastim (G-CSF), sargramostim (GM-CSF), and epoetin alfa for 13 days. Expanded PBMNC are reinfused on day 0.

Patients are followed monthly for 1 year.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven relapsed or refractory non-Hodgkin's lymphoma
* Scheduled to undergo high-dose chemotherapy (carmustine, etoposide, cytarabine, and melphalan) with autologous peripheral blood mononuclear cell transplantation
* No metastatic disease involving the bone marrow

PATIENT CHARACTERISTICS:

Age:

* 17 to 65

Performance status:

* ECOG 0 or 1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* No active hepatitis B or C
* Bilirubin less than 2.5 times normal*
* SGOT or SGPT less than 2.5 times normal*
* Alkaline phosphatase less than 2.5 times normal NOTE: * Unless Gilbert's syndrome present

Renal:

* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* Cardiac ejection fraction normal

Pulmonary:

* DLCO at least 50% predicted
* FEV_1 and FVC at least 75% predicted

Other:

* HIV negative
* Not pregnant
* Negative pregnancy test
* No non-neoplastic disease that would preclude intensive chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior external beam radiotherapy to more than 25% of the active bone marrow

Surgery:

* Not specified

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 1999-09; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane N. Winter, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States